CLINICAL TRIAL: NCT06777056
Title: Artificial Intelligence in the Identification of Lung Contusions Through Chest Radiological Examination in Blunt Thoracic Trauma
Brief Title: AI in the Identification of Lung Contusions Through Chest Radiological Examination in Blunt Thoracic Trauma
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LUNIT
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Lung Contusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The observational study focuses on comparing the interpretation of chest radiological examinations performed using a computer-based system with the standard interpretation conducted by a radiologist. The "LUNIT" system serves as a tool designed to assist radiologists in detecting the 10 most common abnormalities visible on chest radiographs, with proven efficacy in large case series.

The investigation addresses the need to evaluate lung injuries resulting from thoracic trauma, which are linked to a higher risk of complications requiring close monitoring to detect potential respiratory failure.

The primary aim of the study is to assess the accuracy of the LUNIT system in interpreting chest radiographs for the identification of lung contusions compared to the standard radiologist-based interpretation.

DETAILED DESCRIPTION:
The study is observational, cross-sectional, retrospective, and involves a post-marketing device (LUNIT INSIGHT CXR, CE-marked), with a non-profit framework. Patients presenting to the general Emergency Department (ED) of the IRCCS AOU of Bologna with blunt thoracic trauma, who underwent a chest HRCT within 48 hours of a standard chest X-ray, between June 1, 2014, and June 1, 2024, will be retrospectively included. Enrollment will be consecutive and based on discharge reports from the ED.

Chest X-rays will be analyzed using LUNIT by two expert radiologists. The identification of contusions by LUNIT will be compared with the standard chest X-ray reading (based on reports issued at the time of ED presentation), using chest HRCT as the gold standard. No changes will be made to the routine diagnostic-therapeutic pathway of patients. The Radiology Unit involved will be the Radiology Department of IRCCS AOUBO, Policlinico di Sant'Orsola; activities performed by the radiologists will include image reading, interpretation, and reporting, as per standard clinical practice, both before and after the application of LUNIT.

The identification of pulmonary contusions is crucial in the assessment of patients with blunt thoracic trauma, as it significantly impacts clinical management, often necessitating clinical observation due to the risk of respiratory failure and bacterial superinfection. Accurate identification of contusions on chest X-rays can reduce the need for HRCT in high-risk patients.

The use of software like LUNIT could represent a valid alternative to HRCT for patients presenting to the ED with blunt thoracic trauma, potentially reducing ionizing radiation exposure and shortening ED management times. Patients presenting to the general ED of IRCCS AOU of Bologna with blunt thoracic trauma and undergoing HRCT within 48 hours of a chest X-ray between June 1, 2014, and June 1, 2024, will be retrospectively included.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients presenting to the general Emergency Department of the IRCCS AOU of Bologna between June 1, 2014, and June 1, 2024, for blunt thoracic trauma
* Performance of chest HRCT within 48 hours of standard chest X-ray

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department of the IRCCS AOU of Bologna between June 1, 2014, and June 1, 2024, for blunt thoracic trauma, with chest HRCT performed within 48 hours of the chest X-ray.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of lung contusion detection on chest X-rays, with LUNIT software | through study completion, an average of 1 year
  Sensitivity of lung contusion detection on chest X-rays, with and without the use of LUNIT software, compared to the gold standard: chest HRCT performed within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Salvatore, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No